CLINICAL TRIAL: NCT01023126
Title: Poor Patients Adherence to Exercise and Group Therapy as an Approach to Obesity Treatment
Brief Title: Obesity and Psychotherapy as an Alternative to Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feevale (Other)
Responsible Party: Cesar Luis Reichert, Centro Universitario Feevale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 972833
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Obesity; Therapy
Keywords: Obesity; Exercise; Psychotherapy
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EO (No Intervention): Exercise three times a week, one under supervision and two freely chosen by the participant
- EGT (Experimental): Exercise three times a week, one under supervision and two freely chosen by the participant
  Interventions: Behavioral: Group Psychotherapy

INTERVENTIONS:
Behavioral: Group Psychotherapy — Group psychotherapy once a week, under a psychiatrist supervision
  Arms: EGT

SUMMARY:
Adherence to obesity treatment programs has been a limiting factor to good results in loosing weight. This study aimed to verify if obese subjects submitted to a physical exercise program and group psychotherapy would have a greater adherence, than obese people exercising only.

DETAILED DESCRIPTION:
The sample was forty people, both genders, mean age: 42,2 ± 10,7 years old. Physical exercise consisted of walking and stretching three times a week, during 50 minutes, with intensity verified by the Borg Scale, during three months. One of the days were supervised by the authors while two were freely chosen by the participant, without supervision. The verified variables were: total body mass, height, body mass index, physical activity level, caloric expenditure, waist circumference and fat percentile. Half of the sample participated of group psychotherapy once weekly.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 30 kg/m2

Exclusion Criteria:

* Age less than 25 or more than 62

Ages: 25 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Weight loose | three months

CONTACTS AND LOCATIONS:
Overall Officials: Cesar L Reichert, PhD MD, Principal Investigator — Centro Universitário Feevale
Locations (1):
- Centro Universirário Feevale, Novo Hamburgo, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Centro Universitário Feevale webpage — http://www.feevale.br